CLINICAL TRIAL: NCT06610201
Title: Velora Discover: A Prospective, Screening Study of Bleeding and Treatment in Participants With Von Willebrand Disease
Brief Title: A Study of Bleeding and Treatment in Participants With Von Willebrand Disease
Status: Recruiting | Type: Observational
Sponsor: Hemab ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: HMB-002-101_SCR
Record Dates: First submitted 2024-09-13; First posted 2024-09-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Von Willebrand Disease (VWD); Von Willebrand Disease (VWD), Type 1; Von Willebrand Disease (VWD), Type 2; Von Willebrand Disease (VWD), Type 3; Von Willebrand Disease, Type 2A; Von Willebrand Disease, Type 2M; Von Willebrand Disease, Type 2N
Keywords: Von Willebrand Disease (VWD); Prospective Study; Type 1 VWD; Type 2 VWD; Type 3 VWD; Prophylaxis; Von Willebrand Factor (VWF)
MeSH Terms: conditions — von Willebrand Diseases; von Willebrand Disease, Type 2; von Willebrand Disease, Type 3 | interventions — Sarcoglycans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VWD Type 1 (residual VWF antigen and/or activity less than 30 IU per dL)
  Interventions: Other: Clinical outcomes of patients with VWD, Type 1
- VWD Type 2A, Type 2M, Type 2N, or Type 3
  Interventions: Other: Clinical outcomes of patients with VWD, Type 2A, Type 2M, Type 2N, or Type 3

INTERVENTIONS:
Other: Clinical outcomes of patients with VWD, Type 1 — Accumulate information regarding bleeding events, quality of life, and the social and clinical impact of bleeding events in participants with VWD, Type 1
  Groups: VWD Type 1 (residual VWF antigen and/or activity less than 30 IU per dL)
Other: Clinical outcomes of patients with VWD, Type 2A, Type 2M, Type 2N, or Type 3 — Accumulate information regarding bleeding events, quality of life, and the social and clinical impact of bleeding events in participants with VWD, Type 2A, Type 2M, Type 2N and Type 3.
  Groups: VWD Type 2A, Type 2M, Type 2N, or Type 3

SUMMARY:
The purpose of this screening study is to accumulate information regarding bleeding events, quality of life, and the social and clinical impact of bleeds in participants with Von Willebrand Disease (VWD). Data from this study will be used to establish baseline bleeding and treatment rates in a population of participants with VWD and act as comparator data for future clinical study outcomes.(e.g. Velora Pioneer)

DETAILED DESCRIPTION:
This is a prospective, screening study in participants with confirmed Type 1 VWD according to diagnostic guidelines. Participants with confirmed Type 1 VWD and associated bleeding symptoms will be enrolled. The study may also be opened to participants with Type 2 and Type 3 VWD with Sponsor approval. Up to a total of 200 participants may be enrolled in the study.

The study includes screening, a baseline evaluation, and an approximately 4 month observation period which will include every other week telemedicine check-ins (to monitor bleed diary entries and bleeding event treatments. There will be an optional extension to the observation period of up to a total of 12 months for participants wishing to continue.

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to provide informed consent to participate in the study, in accordance with applicable regulations.
2. Has an understanding, ability, and willingness to comply with Study procedures and restrictions.
3. ≥ 16 years at the time of screening.
4. Has congenital Type 1 VWD with a residual VWF antigen and/or activity <30 IU/dL and/or meets the bleeding event rate inclusion criteria. Other congenital VWD subtypes may be enrolled with Sponsor approval.
5. Has symptomatic disease as defined by a history of bruising or bleeding events, with an expected minimum of 3 bleeding episodes (including heavy menstrual bleeding) per year that require treatment to control bleeding symptoms, and/or has recurrent and ongoing episodes of heavy menstrual bleeding at the time of enrollment.

Exclusion Criteria:

1. Has a personal history of venous or arterial thrombosis or thromboembolic disease, except for catheter-associated, superficial vein thrombosis events.
2. Has a significant family history of unprovoked thromboembolic events in first degree relatives.
3. Has a congenital or acquired bleeding disorder other than VWD.
4. Has planned major surgery within the next 6 months.
5. Is pregnant or plans to become pregnant within the next 6 months.
6. Has any concurrent disease, treatment (including ongoing anticoagulation, antiplatelet, or non-steroidal anti-inflammatory drugs), condition, medication, or abnormality in clinical laboratory tests which may impact on the participant's bleeding symptoms or affect their ability to complete the study, in the Investigator's opinion.
7. Has received any investigational product within 30 days prior to screening. If the participant was enrolled and dosed in Velora Pioneer (study HMB-002-102; NCT06754852), they must have completed their End of Study Visit.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants ≥16 years of age with VWD.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding event rate | 4.5 to 12.5 months
Annualized treated bleeding rate | 4.5 to 12.5 months
Annualized heavy menstrual bleed rate | 4.5 to 12.5 months
Number of overnight admissions | 4.5 to 12.5 months
  Hospitalization monitoring of bleeding events.

SECONDARY OUTCOMES:
Prophylactic and on demand treatment | 4.5 to 12.5 months
  Details of treatment used for bleeding events
Iron status | 4.5 to 12.5 months
  Blood samples will be collected for the determination of ferritin and hemoglobin.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 | 4.5 to 12.5 months
  An assessment which evaluates four items from each of the seven PROMIS domains. Each question is rated on a scale of 1 to 5. In addition, the PROMIS-29 includes one pain intensity question which is rated on a scale of 1 to 10. Higher scores on the PROMIS-29 indicate worse symptoms.
Menstrual Bleeding Questionnaire (MBQ) | 4.5 to 12.5 months
  Measure the effect of heavy menstrual bleeding on a self-assessment of menstrual blood loss, limitations in social and leisure activities, physical activities, and work activities.
Epistaxis Severity Score (ESS) | 4.5 to 12.5 months
  Assessment of nose bleed severity
Oral Bleeding Experience | 4.5 to 12.5 months
  Questionnaire to evaluate bleeding symptoms

CONTACTS AND LOCATIONS:
Overall Officials: VP of Clinical Research, Study Director — Hemab ApS
Locations (17):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Miami Hospital and Clinics, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Innovative Hematology, Inc./Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Michigan Hospitals, Department of Hemophilia and Coagulation Disorders, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Washington Institute For Coagulation (WIC), Seattle, Washington
- Australia (3):
  - Fiona Stanley Hospital, Murdoch, Perth
  - Royal Prince Alfred Hospital, Camperdown, Sydney
  - The Alfred Hospital, Melbourne, Victoria
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No